CLINICAL TRIAL: NCT04242329
Title: Surgery of Melanoma Metastases After Systemic Therapy - the SUMMIST Trial
Brief Title: Surgery of Melanoma Metastases After Systemic Therapy
Acronym: SUMMIST
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not possible to recruit patients during COVID, and not possible to start enrolling after the pandemic.
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Associate professor, Senior Consultant Surgeon, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUMMIST
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Melanoma; Melanoma Stage IV; Metastatic Melanoma; Surgery
Keywords: Immunotherapy; Metastatic surgery; Surgical oncology
MeSH Terms: conditions — Melanoma | interventions — Immunotherapy

STUDY DESIGN:
Intervention Model Description: A Phase II Randomized Controlled Open-Label Parallel Group Interventional Multicenter Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD1-inhibitor + surgery (Experimental): Patients randomised to the interventional study arm, receiving both surgical metastasectomy and continued immunotherapy. Each patient case will be individually planned for surgery. Procedures will include, but will not be limited to, lung resections, liver resections, bowel resection, skin excisions and lymph node clearances. Patients in both study arms will continue with PD-1 inhibitor 12 months after randomization, and will then be treated according to their medical oncologist.
  Interventions: Procedure: Surgical metastasectomy
- PD1-inhibitor (Active Comparator): Patients randomized to control study arm, receiving continued immunotherapy only. Patients in both study arms will continue with PD-1 inhibitor 12 months after randomization, and will then be treated according to their medical oncologist.
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Procedure: Surgical metastasectomy — Surgical removal of metastases aimed at R0 resection.
  Arms: PD1-inhibitor + surgery
Drug: Immunotherapy — Continued PD1-inhibitor treatment according to current treatment standards.
  Arms: PD1-inhibitor

SUMMARY:
To evaluate if surgical removal of residual disease adds benefit in stage IV melanoma patients with partial response or stable disease after a minimum 9 months of first-line PD-1 inhibition. Primary endpoint: Disease-free survival (DFS) at 12 months.

DETAILED DESCRIPTION:
A Phase II Randomized Controlled Open-Label Parallel Group Interventional Multicenter Trial. Patients with metastatic melanoma, stratified for stage M1a or M1b/M1c, that have received first-line treatment with PD-1 inhibitors for a minimum of 9 months resulting in either partial response or stable disease according to RECIST 1.1 will be eligible. Patients will be screened for operability based on CT-scans examined by a multidisciplinary team, with the criteria that complete (R0) resection of all metastases should be possible. If the multidisciplinary team find that this would be possible, patients will be included and randomized 1:1 to either surgery with continued PD1-inhibition or current standard of care with continued PD1-inhibition only. At progression, treatment will be according to the treating medical oncologist. Active follow-up will be performed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Signed and dated written informed consent before the start of specific protocol procedures
* Biopsy or cytology proven metastatic melanoma stage M1a, M1b or M1c
* Have received a minimum of 9 months of immunotherapy (PD1-inhibitor alone or in combination) resulting in stable disease or partial response according to RECIST 1.1
* Metastases judged to be radically resectable by surgery at a multidisciplinary conference
* ECOG performance status 0-2

Exclusion Criteria:

* Brain metastasis (M1d)
* Previous treatment with BRAF/MEK inhibitors
* Inability to understand given information or undergo study procedures according to protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
DFS 12 months | 12 months
  Disease free survival

SECONDARY OUTCOMES:
SAE 12 months | 12 months
  Serious adverse events
Complications | 3 months post operatively
  Surgical complications according to the Clavien-Dindo classification
R0 resection | 3 months post operatively
  Rate of R0 resections according to pathology report
PFS 12 months | 12 months
  Progression free survival
MSS 12 months | 12 months
  Melanoma specific survival
OS 12 months | 12 months
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No